CLINICAL TRIAL: NCT07271433
Title: Continuous Glucose Monitoring for Post-kidney Transplantation in Pre-existing Type 2 Diabetes
Status: Active, not recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 23-390
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Kidney Transplant
Keywords: CGM; Kidney Transplant; Continuous Glucose Monitor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post Kidney Transplant, using CGM: A total of 20 patients that are post kidney transplant, will wear a Continuous Glucose Monitor (CGM) until 3 months post-transplant.

SUMMARY:
Use of continuous glucose monitor (CGM) in post kidney transplant patients to better assess changes in glucose levels post kidney transplant

DETAILED DESCRIPTION:
This is a non-randomized perspective single arm study with a planned enrollment of 20 patients. The primary objective is to characterize the glucometrics (description of glucose readings in relation to target goals) achieved by a CGM-based insulin titrating protocol for glucocorticoid taper for post kidney transplant patients. The secondary objective is to explore the relationship between the CGM glucometrics and rates of readmission, rejection and delayed graft function in post kidney transplant patients.

A total of 20 patients that are post kidney transplant, will undergo intervention until 3 months post-transplant. Informed consent will be obtained prior to start of study. The final visit will be at 3 months. Patients will be discharged to their local endocrinologist or primary care physician at this 3-month mark. Data will continue to be gathered for 3 more months after exit from intervention. Enrollment will be within the first 2 weeks of hospital discharge. Visits are standard of care (SOC) at the Kidney Transplant Clinic or at the Endocrinology clinic and will be virtual, in-person or telephone encounter.

ELIGIBILITY:
Inclusion Criteria:

1. Sex: men and women
2. Ethnicity: all ethnic groups
3. Age: ≥ 18
4. Known type 2 diabetes before kidney transplant
5. Kidney transplant alone
6. On multiple daily insulin injection
7. Standard prednisone taper
8. Smart phone - compatible with the LibreView App

Exclusion Criteria:

1. Simultaneous pancreas-kidney transplant
2. Allergy to Freestyle Libre components including adhesive
3. Use of vitamin C at doses 500 mg or greater
4. Blood dyscrasias that prevent hemoglobin A1c interpretation
5. Lack of mobile app accessibility
6. Rapid prednisone taper

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a non-randomized prospective single arm study with a planned enrollment of 20 patients.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Time in Range (TIR) | 6 months
  Percent of patients who achieved Time in Range (55 mg/dL to 180 mg/dL Glucose) as measured by the Continuous Glucose Monitor
Hospital Readmission | 6 months
  Percent of patients who experienced a hospital readmission
Time below range (TBR) | 6 months
  Percent of patients who achieved Time below range (<54 mg/dL Glucose) as measured by the Continuous Glucose Monitor
Time above range (TAR) | 6 months
  Percent of patients who achieved Time above range (181-250mg/dL and >250 mg/dL Glucose) as measured by the Continuous Glucose Monitor
Rejection | 6 months
  Percent of patients who experienced a rejection of the transplanted kidney
Delayed graft function | 6 months
  Percent of patients who experienced delayed graft function

CONTACTS AND LOCATIONS:
Locations (1):
- The Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to the disclosure on the consent form for which IRB approval was received. Deidentified summarized results will be shared via publication in a medical journal

DOCUMENTS (1):
  • Study Protocol (2024-06-24): https://cdn.clinicaltrials.gov/large-docs/33/NCT07271433/Prot_000.pdf